CLINICAL TRIAL: NCT05455632
Title: Can Postoperative Radiotherapy be Omitted for Oral Squamous Cell Carcinoma Patients Underwent Neoadjuvant Therapy and Surgery? - A Retrospective Cohort Study
Brief Title: Postoperative Radiotherapy for Oral Squamous Cell Carcinoma After Neoadjuvant Therapy and Surgery
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: PORT-NAT
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Radiotherapy; Neoadjuvant Therapy; Oral Squamous Cell Carcinoma; Surgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1:PORT: Oral squamous cell carcinoma (OSCC) patients received neoadjuvant therapy, surgery, and postoperative radiotherapy.
- Group2:non-PORT: Oral squamous cell carcinoma (OSCC) patients received neoadjuvant therapy and surgery, without postoperative radiotherapy

SUMMARY:
The treatment guideline for locally advanced resectable oral squamous cell carcinoma (LAROSCC) is surgery + postoperative radiotherapy/chemoradiotherapy. Though the treatment is intensive with serious harm to quality of life, the survival of patients is poor. Neoadjuvant therapy has been evaluated in a number of clinical trials for LAROSCC, but failed to directly improve the overall survival. On the other hand, de-escalation of treatment followed by neoadjuvant is also been explored with some promising results. This study is to retrospectively include patients with LAROSCC who received neoadjuvant therapy and surgery. Survival between patients in two cohorts (cohort 1: received postoperative radiotherapy, cohort 2: received no postoperative radiotherapy) are to be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving neoadjuvant therapy and surgery for oral squamous cell carcinoma from January 2008 to December 2021
* Oral squamous cell carcinoma histology (including tongue, gingiva, cheek, floor of mouth, hard palate and posterior molar area)
* Clinical stage III/IVA (T1-2/N1-2/M0 or T3-4/cN0-2/M0, AJCC 2018) for the primary lesion
* Surgical resection samples that can be evaluated for pathological remission rate

Exclusion Criteria:

* Severe/active systemic disease
* Previously radiotherapy or neck lymph node dissection for the head and neck region
* Evidence of tumor recurrence or metastasis in physical examination or imaging (ultrasound, CT, MRI) before initiation adjuvant radiotherapy
* Evidence of severe/unrelieved side effects of neoadjuvant therapy or severe postoperative complications before initiation adjuvant radiotherapy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Oral squamous cell carcinoma (OSCC) patients received neoadjuvant therapy and surgery with and without postoperative radiotherapy in the Department of Oral and Maxillofacial-Head and Neck Oncology in Ninth People's Hospital, Shanghai JiaoTong University School of Medicine from January 2008 to December 2021.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
OS | 24 months
  Overall survival

SECONDARY OUTCOMES:
LRFS | 24 months
  Local recurrence-free rate
QOL | 24 months
  Quality of life (QOL), according to the QLQ-C30 scoring manual, the final QOL scores of each field are transformed into standardized scores within 0-100 through linear transformation
OS-MPR | 24 months
  Overall survival for patients obtained major pathological response (MPR) from neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, Principal Investigator — Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ju W, Zhang Y, Liu Y, Sun J, Li J, Dong M, Sun Q, Shi W, Zhao T, Zhou Z, Huang Y, Zhou X, Zhu D, Dou S, Zhang Z, He Y, Zhang C, Xia R, Zhu G, Zhong L. Can adjuvant radiotherapy be omitted for oral cavity cancer patients who received neoadjuvant therapy and surgery? A retrospective cohort study. Int J Surg. 2023 Apr 1;109(4):879-886. doi: 10.1097/JS9.0000000000000353. PMID 36999830